CLINICAL TRIAL: NCT04555889
Title: The Impact of Lung Recruitment Maneuver in 24-32 Weeks Preterm Babies With Assist-control Volume Guarantee Mode to Their Hemodynamic Status and the Incidence of Bronchopulmonary Dysplasia
Brief Title: The Impact of Lung Recruitment Maneuver in 24-32 Weekers, and the Incidence of Bronchopulmonary Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. R. Adhi Teguh Perma Iskandar, Sp.A(K) (Other)
Collaborators: Indonesia Medical Education and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. R. Adhi Teguh Perma Iskandar, Sp.A(K), Principal Investigator of Perinatology Division, Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Med. Fac. of Univ. Indonesia
Record Dates: First submitted 2020-08-12; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: lung recruitment maneuver; preterm babies; Bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: The impact of lung recruitment maneuver in 24-32 weekers with assist-control volume guarantee mode to their hemodynamic status and the incidence of Bronchopulmonary dysplasia
Who Masked: Participant, Outcomes Assessor
Masking Description: * All babies wether they experience the intervention ofr not they can not tell to other peoples.
  * Only The lab analyzer will be blind to the subject of study, other measurement can not be blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lung recruitment maneuver (LRM) group (Experimental): The lung recruitment maneuver (LRM) will be done by increasing of PEEP 0,2 cm H2O every 3 minutes, until reach the opening pressure. After that PEEP decrease gradually until get the closing pressure. Than the investigators will back to the opening pressure for 3 minutes, and the final PEEP will be put backo 0,2 above closing pressure.
  Interventions: Device: lung recruitment maneuver (LRM) with DrageerVN500
- without lung recruitment maneuver (LRM) group (No Intervention): Another group get standart protocol only.

INTERVENTIONS:
Device: lung recruitment maneuver (LRM) with DrageerVN500 — interventions involving device that may help to gradually lung development
  Arms: lung recruitment maneuver (LRM) group

SUMMARY:
hypothesis :

1. The incident of dysplasia bronchopulmonary and/or death in 24-32 weekers babies on assist-control volume guarantee ventilation are lower in lung recruitment maneuver (LRM) group compare to control.
2. The serum levels of surfactant protein-D in 24-32 weekers babies on assist-control volume guarantee ventilation are lower in lung recruitment maneuver (LRM) group compare to control.
3. The serum concentration of CD-31+ and CD-42b- in 24-32 weekers babies on assist-control volume guarantee ventilation are lower in lung recruitment maneuver (LRM) group compare to control.
4. The right and left cardiac output in 24-32 weekers babies on assist-control volume guarantee mode are more higher in lung recruitment maneuver (LRM) group, than group that did not get LRM
5. The incident Patent Ductus Arteriosus in 24-32 weekers babies on assist-control volume guarantee ventilation are lower in lung recruitment maneuver (LRM) group compare to control.
6. The difference tc-pCO2 - PaCO2 , tcO2 index , and strong ion difference (SID) in 24-32 weekers babies on assist-control volume guarantee ventilation are lower in lung recruitment maneuver (LRM) group compare to control.

DETAILED DESCRIPTION:
description of the protocol :

1. All Babies that meet inclusion criteria would immediately given surfactan. Babies will do echocardiography, blood gas analize, blood sample, transcutaneous monitor. After that babies will be randomized, the intervention group will get standart protocol + lung recruitment maneuver (LRM) and another group get standart protocol only.
2. The lung recruitment maneuver (LRM) will be done by increasing of PEEP 0,2 cm H2O every 3 minutes, until reach the opening pressure. After that PEEP decrease gradually until get the closing pressure. Than the investigators will back to the opening pressure for 3 minutes, and the final PEEP will be put back 0,2 above closing pressure.
3. After 3rd days (72 hours) babies, the investigators will exime serum levels of surfactan protein-D, CD-31+ and CD-42b- , blood gas , tc-pCO2 - PaCO2 , tcO2 index.
4. After that babies will observe within 28 days to detect Bronchopulmonary dysplasia

ELIGIBILITY:
Inclusion Criteria:

* 24-32 weeks preterm babies.
* Babies on assist-control volume guarantee ventilation with FiO2 > 30% to reach oxygen saturations within 90-95%.
* Age less than 48 hours.
* Born in Cipto Mangunkusumo Hospital and Bunda Menteng Hospital.
* Parents/guardians agreed to participate in this study with sign informed consent.

Exclusion Criteria:

* Weight birth <750 grams.
* APGAR score at 10 minutes are <5.
* Born with congenital heart disease except patent ductus arteriosus or presistence foramen ovale.
* Born with congenital disorder that need surgery intervention (for example :

diaphragmatic hernia, atresia ani, esophageal atresia, duodenal atresia.

* Born with congenital disorder that worsening of the respiratory distress (for example

  * hydrops fetalis, phrenic nerve paralysis, abnormality of chest wall, abnormality of air way (for example : Choanal atresia, Laryngeal stenosis, cleft palate.
* Born inborn error metabolism disease.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowing the relationship between lung recruitment maneuver in 24-32 weeks preterm babies with the incidence of Bronchopulmonary dysplasia | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will have lower incidence of Bronchopulmonary dysplasia compare to control.

SECONDARY OUTCOMES:
Knowing the relationship between lung recruitment maneuver in 24-32 weekers, with their alveolar intergrity (serum levels of surfactan protein-D) | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will have lower serum levels of surfactan protein -D compare to control.
Knowing the relationship between lung recruitment maneuver in 24-32 weekers, with their lung endothel intergrity (serum levels of CD-31+) | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will have lower serum concentrarion of CD-31+ compare to control.
Knowing the relationship between lung recruitment maneuver in 24-32 weeks preterm babies with their lung endothel intergrity (serum levels of CD-42b-) | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will have lower serum concentrarion of CD-42b- compare to control.
Knowing the relationship between lung recruitment maneuver in 24-32 weeks preterm babies with their micro circulation (oxygen index) | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will have higher oxygen index compare to control.
Knowing the relationship between lung recruitment maneuver in 24-32 weeks preterm babies with their their micro circulation (tc-pCO2 - PaCO2 index) | 12 weeks
  preterm babies ( 24-32 weeks) with Lung Recrutment manuver will have transcutaneous-arterial partial carbon dioxide gap lower than control ( less than 6 mmHg ). babies with better microcirculation status will show less than 6 mmHg transcutaneous-arterial partial carbon dioxide gap.
Knowing the relationship between lung recruitment maneuver in 24-32 weeks preterm babies with their incidence patent ductus arteriosus (PDA) significant | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will make lower incident of Patent Ductus Arteriosus compare to control.
Knowing the relationship between lung recruitment maneuver in 24-32 weeks preterm babies with their macro circulation | 12 weeks
  Preterm babies ( 24-32 weeks) with Lung Recruitment maneuver will make right and left cardiac output higher compare to control.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. R. Adhi T Perma Iskandar, Sp.A (K), Principal Investigator — RSCMPerinatology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Result] Liu L, Oza S, Hogan D, Chu Y, Perin J, Zhu J, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of under-5 mortality in 2000-15: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet. 2016 Dec 17;388(10063):3027-3035. doi: 10.1016/S0140-6736(16)31593-8. Epub 2016 Nov 11. PMID 27839855
- [Result] Kumar A, Bhat BV. Epidemiology of respiratory distress of newborns. Indian J Pediatr. 1996 Jan-Feb;63(1):93-8. doi: 10.1007/BF02823875. PMID 10829971
- [Result] van Kaam AH, de Jaegere A, Haitsma JJ, Van Aalderen WM, Kok JH, Lachmann B. Positive pressure ventilation with the open lung concept optimizes gas exchange and reduces ventilator-induced lung injury in newborn piglets. Pediatr Res. 2003 Feb;53(2):245-53. doi: 10.1203/01.PDR.0000047520.44168.22. PMID 12538782
- [Result] Peng W, Zhu H, Shi H, Liu E. Volume-targeted ventilation is more suitable than pressure-limited ventilation for preterm infants: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F158-65. doi: 10.1136/archdischild-2013-304613. Epub 2013 Nov 25. PMID 24277660
- [Result] DiBlasi RM. Neonatal noninvasive ventilation techniques: do we really need to intubate? Respir Care. 2011 Sep;56(9):1273-94; discussion 1295-7. doi: 10.4187/respcare.01376. PMID 21944681
- [Result] Haczku A. Protective role of the lung collectins surfactant protein A and surfactant protein D in airway inflammation. J Allergy Clin Immunol. 2008 Nov;122(5):861-79; quiz 880-1. doi: 10.1016/j.jaci.2008.10.014. PMID 19000577
- [Result] Eisner MD, Parsons P, Matthay MA, Ware L, Greene K; Acute Respiratory Distress Syndrome Network. Plasma surfactant protein levels and clinical outcomes in patients with acute lung injury. Thorax. 2003 Nov;58(11):983-8. doi: 10.1136/thorax.58.11.983. PMID 14586055
- [Result] Reid VL, Webster NR. Role of microparticles in sepsis. Br J Anaesth. 2012 Oct;109(4):503-13. doi: 10.1093/bja/aes321. Epub 2012 Sep 4. PMID 22952169
- [Result] Woodfin A, Voisin MB, Nourshargh S. PECAM-1: a multi-functional molecule in inflammation and vascular biology. Arterioscler Thromb Vasc Biol. 2007 Dec;27(12):2514-23. doi: 10.1161/ATVBAHA.107.151456. Epub 2007 Sep 13. PMID 17872453
- [Result] Cabrera-Benitez NE, Valladares F, Garcia-Hernandez S, Ramos-Nuez A, Martin-Barrasa JL, Martinez-Saavedra MT, Rodriguez-Gallego C, Muros M, Flores C, Liu M, Slutsky AS, Villar J. Altered Profile of Circulating Endothelial-Derived Microparticles in Ventilator-Induced Lung Injury. Crit Care Med. 2015 Dec;43(12):e551-9. doi: 10.1097/CCM.0000000000001280. PMID 26308427
- [Result] Kluckow M, Evans N. Superior vena cava flow in newborn infants: a novel marker of systemic blood flow. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F182-7. doi: 10.1136/fn.82.3.f182. PMID 10794783
- [Result] Bancalari E, Claure N. Definitions and diagnostic criteria for bronchopulmonary dysplasia. Semin Perinatol. 2006 Aug;30(4):164-70. doi: 10.1053/j.semperi.2006.05.002. PMID 16860155
- [Result] Madurga A, Mizikova I, Ruiz-Camp J, Morty RE. Recent advances in late lung development and the pathogenesis of bronchopulmonary dysplasia. Am J Physiol Lung Cell Mol Physiol. 2013 Dec;305(12):L893-905. doi: 10.1152/ajplung.00267.2013. Epub 2013 Nov 8. PMID 24213917
- [Result] Castoldi F, Daniele I, Fontana P, Cavigioli F, Lupo E, Lista G. Lung recruitment maneuver during volume guarantee ventilation of preterm infants with acute respiratory distress syndrome. Am J Perinatol. 2011 Aug;28(7):521-8. doi: 10.1055/s-0031-1272970. Epub 2011 Mar 4. PMID 21380992
- See also: Heated, humidified high-flow nasal cannula vs. nasal CPAP in infants with moderate respiratory distress — https://www.paediatricaindonesiana.org/index.php/paediatrica-indonesiana/article/view/2203
- See also: Experimental Ventilator-induced Lung Injury: Exacerbation by Positive End-Expiratory Pressure — https://pubs.asahq.org/anesthesiology/article/110/6/1341/10637/Experimental-Ventilator-induced-Lung
- See also: Transitional Hemodynamics in Preterm Neonates: Clinical Relevance — https://doi.org/10.1016/j.pedneo.2015.07.002